CLINICAL TRIAL: NCT00360893
Title: Epidemiology of Diabetes Interventions and Complications (EDIC)
Status: Active, not recruiting | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: N01-DK-6-2204; U01DK094176 (NIH)
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Diabetes Control and Complications Trial (DCCT,1983-1993) compared intensive therapy aimed at near-normal glycemia versus conventional therapy with no specific glucose targets in 1441 subjects with type 1 diabetes (T1DM) over a mean follow-up of 6.5 years. Intensive therapy reduced the risks of retinopathy, nephropathy, and neuropathy by 35-76%. The level of glycemia was the primary determinant of complications. We also described the adverse effects of intensive therapy; assessed its effects on cardiovascular disease (CVD) risk factors, neurocognition and quality of life; and projected the lifetime health-economic impact. After the primary DCCT results were reported in 1993, intensive therapy aiming for a HbA1c <7% was adopted world-wide as standard-of-care for T1DM.

The Epidemiology of Diabetes Interventions and Complications (EDIC, 1994-present) is the observational follow-up study of the DCCT cohort. Micro- and cardio-vascular complications and a wide range of established and putative risk factors, including genetic and epigenetic factors, have been measured with standardized methods, carefully documented and events adjudicated. EDIC has notably shown that the early beneficial effects of intensive versus conventional therapy on complications persisted for ~15 years despite the convergence of HbA1c levels in the two groups during EDIC, a novel concept termed metabolic memory. Prior intensive therapy was also shown to reduce substantially the risk of CVD events and mortality.

The overarching goals for the current cycle (2022-2027) are to study the occurrence and identify potentially modifiable risk factors of the more advanced microvascular and cardiovascular complications and physical and cognitive dysfunction that are occurring with increasing diabetes duration and age. With increasing longevity, the increased adiposity that has affected patients with T1DM, including EDIC participants, has potential adverse consequences. Thus, the impact of diabetes duration, aging and adiposity on morbidities and their underlying risk factors will be studied. The results will guide treatment priorities as T1DM patients age.

ELIGIBILITY:
Participants originally enrolled in the Diabetes Control and Complications Trial (DCCT) (N01-DK-6-2204-A).

Ages: 19 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Participants originally enrolled in the Diabetes Control and Complications Trial (DCCT) (N01-DK-6-2204-A).
Sampling Method: Non-Probability Sample
Enrollment: 1441 (Actual)
Dates: Start 1994-04; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
2022-2027 Cycle | Eyes (Yrs 32-33, 2025-26); Kidney (annually); Nerves (Yrs 29-31, 33-34, 2022-26); CVD events (continuous, adjudicated annually); Physical (Yrs 29-31, 2022-24); Cognitive (Yrs 32-33, 2025-26); Liver (Yrs 29-31, 2022-24); Sleep (Yrs 29-31, 2022-24).
  Advanced microvascular complications (retinopathy, kidney disease, neuropathy), major CVD events or early subclinical, changes in physical and cognitive dysfunction, fibrosis and steatosis, obstructive sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: David M Nathan, M.D., Study Chair — Massachusetts General Hospital; Rose A Gugitosi-Klug, M.D., Ph.D., Principal Investigator — Case Western Reserve University; Barbara H Braffett, Ph.D., Principal Investigator — George Washington University; Ionut Bebu, Ph.D., Principal Investigator — George Washington University

IPD SHARING:
Plan to Share IPD: Yes
NIDDK Central Repository

REFERENCES:
- [Result] DCCT/EDIC Research Group; Nathan DM, Bebu I, Hainsworth D, Klein R, Tamborlane W, Lorenzi G, Gubitosi-Klug R, Lachin JM. Frequency of Evidence-Based Screening for Retinopathy in Type 1 Diabetes. N Engl J Med. 2017 Apr 20;376(16):1507-1516. doi: 10.1056/NEJMoa1612836. PMID 28423305
- [Result] Writing Group for the DCCT/EDIC Research Group; Orchard TJ, Nathan DM, Zinman B, Cleary P, Brillon D, Backlund JY, Lachin JM. Association between 7 years of intensive treatment of type 1 diabetes and long-term mortality. JAMA. 2015 Jan 6;313(1):45-53. doi: 10.1001/jama.2014.16107. PMID 25562265
- [Result] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study Research Group; Jacobson AM, Musen G, Ryan CM, Silvers N, Cleary P, Waberski B, Burwood A, Weinger K, Bayless M, Dahms W, Harth J. Long-term effect of diabetes and its treatment on cognitive function. N Engl J Med. 2007 May 3;356(18):1842-52. doi: 10.1056/NEJMoa066397. PMID 17476010
- [Result] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Result] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group; Lachin JM, Genuth S, Cleary P, Davis MD, Nathan DM. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive therapy. N Engl J Med. 2000 Feb 10;342(6):381-9. doi: 10.1056/NEJM200002103420603. PMID 10666428
- [Result] Braffett BH, Bebu I, El Ghormli L, Cowie CC, Sivitz WI, Pop-Busui R, Larkin ME, Gubitosi-Klug RA, Nathan DM, Lachin JM, Dagogo-Jack S; DCCT/EDIC Research Group. Cardiometabolic Risk Factors and Incident Cardiovascular Disease Events in Women vs Men With Type 1 Diabetes. JAMA Netw Open. 2022 Sep 1;5(9):e2230710. doi: 10.1001/jamanetworkopen.2022.30710. PMID 36074461
- [Result] Writing Team for the DCCT/EDIC Research Group; Gubitosi-Klug RA, Sun W, Cleary PA, Braffett BH, Aiello LP, Das A, Tamborlane W, Klein R. Effects of Prior Intensive Insulin Therapy and Risk Factors on Patient-Reported Visual Function Outcomes in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Cohort. JAMA Ophthalmol. 2016 Feb;134(2):137-45. doi: 10.1001/jamaophthalmol.2015.4606. PMID 26584339
- [Result] DCCT/EDIC Research Group; Aiello LP, Sun W, Das A, Gangaputra S, Kiss S, Klein R, Cleary PA, Lachin JM, Nathan DM. Intensive diabetes therapy and ocular surgery in type 1 diabetes. N Engl J Med. 2015 Apr 30;372(18):1722-33. doi: 10.1056/NEJMoa1409463. PMID 25923552
- [Result] DCCT/EDIC Research Group; de Boer IH, Sun W, Cleary PA, Lachin JM, Molitch ME, Steffes MW, Zinman B. Intensive diabetes therapy and glomerular filtration rate in type 1 diabetes. N Engl J Med. 2011 Dec 22;365(25):2366-76. doi: 10.1056/NEJMoa1111732. Epub 2011 Nov 12. PMID 22077236
- [Result] Writing Team for the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Sustained effect of intensive treatment of type 1 diabetes mellitus on development and progression of diabetic nephropathy: the Epidemiology of Diabetes Interventions and Complications (EDIC) study. JAMA. 2003 Oct 22;290(16):2159-67. doi: 10.1001/jama.290.16.2159. PMID 14570951
- [Result] Nathan DM, Lachin J, Cleary P, Orchard T, Brillon DJ, Backlund JY, O'Leary DH, Genuth S; Diabetes Control and Complications Trial; Epidemiology of Diabetes Interventions and Complications Research Group. Intensive diabetes therapy and carotid intima-media thickness in type 1 diabetes mellitus. N Engl J Med. 2003 Jun 5;348(23):2294-303. doi: 10.1056/NEJMoa022314. PMID 12788993
- [Result] Writing Team for the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Effect of intensive therapy on the microvascular complications of type 1 diabetes mellitus. JAMA. 2002 May 15;287(19):2563-9. doi: 10.1001/jama.287.19.2563. PMID 12020338
- [Derived] Rubin M, Kazakia G, Braffett BH, Gregory NS, Lin MH, Trapani V, de Boer IH, Agarwal S, Burghardt A, Guo XE, Gubitosi-Klug R, Schwartz AV; DCCT/EDIC Research Group. Bone microarchitecture assessed by High-resolution peripheral quantitative computed tomography in type 1 diabetes: the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications study. JBMR Plus. 2025 Oct 22;9(12):ziaf167. doi: 10.1093/jbmrpl/ziaf167. eCollection 2025 Dec. PMID 41235023
- [Derived] Braffett BH, El Ghormli L, Martin C, White NH, Hirsch IB, Bantle A, Carlson A, Leschek E, Gubitosi-Klug R, Soliman EZ, Vella A, Perkins BA, Bebu I, Pop-Busui R; DCCT/EDIC Research Group. Cardiovascular autonomic neuropathy defined by indices of heart rate variability is associated with cardiovascular disease: a longitudinal cohort study of participants with type 1 diabetes. Cardiovasc Diabetol. 2025 Aug 13;24(1):334. doi: 10.1186/s12933-025-02856-9. PMID 40804720
- [Derived] Helmink MAG, Hageman SHJ, Visseren FLJ, de Ranitz-Greven WL, de Valk HW, van Sloten TT, Westerink J. Variability in benefit from intensive insulin therapy on cardiovascular events in individuals with type 1 diabetes: A post hoc analysis of the DCCT/EDIC study. Diabet Med. 2023 Nov;40(11):e15183. doi: 10.1111/dme.15183. Epub 2023 Jul 24. PMID 37470718
- [Derived] Khatri M, Ryan CM, Gao X, de Boer IH, Braffett BH, Molitch M, Karger AB, Lorenzi GM, Lee P, Trapani VR, Lachin JM, Jacobson AM. CKD Associates with Cognitive Decline in Middle-Aged and Older Adults with Long-Standing Type 1 Diabetes. Kidney360. 2023 Aug 1;4(8):1058-1071. doi: 10.34067/KID.0000000000000178. Epub 2023 Jun 9. PMID 37291722
- [Derived] Lachin JM, Bebu I, Gao X, Nathan DM, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group. Association of Estimated Time-in-Range Capillary Glucose Levels Versus HbA1c With Progression of Microvascular Complications in the Diabetes Control and Complications Trial. Diabetes Care. 2022 Oct 1;45(10):2445-2448. doi: 10.2337/dc21-2298. PMID 35972222
- [Derived] Martin CL, Trapani VR, Backlund JC, Lee P, Braffett BH, Bebu I, Lachin JM, Jacobson AM, Gubitosi-Klug R, Herman WH; DCCT/EDIC Research Group. Physical Function in Middle-aged and Older Adults With Type 1 Diabetes: Long-term Follow-up of the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study. Diabetes Care. 2022 Sep 1;45(9):2037-2045. doi: 10.2337/dc21-2119. PMID 35880807
- [Derived] Jacobson AM, Braffett BH, Erus G, Ryan CM, Biessels GJ, Luchsinger JA, Bebu I, Gubitosi-Klug RA, Desiderio L, Lorenzi GM, Trapani VR, Lachin JM, Bryan RN, Habes M, Nasrallah IM; DCCT/EDIC Research Group. Brain Structure Among Middle-aged and Older Adults With Long-standing Type 1 Diabetes in the DCCT/EDIC Study. Diabetes Care. 2022 Aug 1;45(8):1779-1787. doi: 10.2337/dc21-2438. PMID 35699949
- [Derived] Gubitosi-Klug RA, Braffett BH, Bebu I, Johnson ML, Farrell K, Kenny D, Trapani VR, Meadema-Mayer L, Soliman EZ, Pop-Busui R, Lachin JM, Bergenstal RM, Tamborlane WV. Continuous Glucose Monitoring in Adults With Type 1 Diabetes With 35 Years Duration From the DCCT/EDIC Study. Diabetes Care. 2022 Mar 1;45(3):659-665. doi: 10.2337/dc21-0629. PMID 35076697
- [Derived] Carlson NE, Horton KW, Hokanson JE, Cleary PA, Jacobs DR Jr, Brunzell JD, Purnell JQ; DCCT/EDIC research group. Weight gain trajectories and obesity rates in intensive and conventional treatments of type 1 diabetes from the DCCT compared with a control population without diabetes. Diabet Med. 2022 May;39(5):e14794. doi: 10.1111/dme.14794. Epub 2022 Jan 26. PMID 35040196
- [Derived] Perkins BA, Bebu I, Gao X, Karger AB, Hirsch IB, Karanchi H, Molitch ME, Zinman B, Lachin JM, de Boer IH. Early Trajectory of Estimated Glomerular Filtration Rate and Long-term Advanced Kidney and Cardiovascular Complications in Type 1 Diabetes. Diabetes Care. 2022 Mar 1;45(3):585-593. doi: 10.2337/dc21-1883. PMID 35015817
- [Derived] Boyko EJ, Zelnick LR, Braffett BH, Pop-Busui R, Cowie CC, Lorenzi GM, Gubitosi-Klug R, Zinman B, de Boer IH. Risk of Foot Ulcer and Lower-Extremity Amputation Among Participants in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study. Diabetes Care. 2022 Feb 1;45(2):357-364. doi: 10.2337/dc21-1816. PMID 35007329
- [Derived] Steigmann L, Miller R, Trapani VR, Giannobile WV, Braffett BH, Pop-Busui R, Lorenzi G, Herman WH, Sarma AV; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Type 1 diabetes and oral health: Findings from the Epidemiology of Diabetes Interventions and Complications (EDIC) study. J Diabetes Complications. 2022 Apr;36(4):108120. doi: 10.1016/j.jdiacomp.2021.108120. Epub 2022 Jan 3. PMID 35000860
- [Derived] Polak JF, Backlund JC, Budoff M, Raskin P, Bebu I, Lachin JM; DCCT/EDIC Research Group. Coronary Artery Disease Events and Carotid Intima-Media Thickness in Type 1 Diabetes in the DCCT/EDIC Cohort. J Am Heart Assoc. 2021 Dec 21;10(24):e022922. doi: 10.1161/JAHA.121.022922. Epub 2021 Dec 7. PMID 34873921
- [Derived] Pop-Busui R, Braffett BH, Wessells H, Herman WH, Martin CL, Jacobson AM, Sarma AV. Diabetic Peripheral Neuropathy and Urological Complications in Type 1 Diabetes: Findings From the Epidemiology of Diabetes Interventions and Complications Study. Diabetes Care. 2022 Jan 1;45(1):119-126. doi: 10.2337/dc21-1276. PMID 34728530
- [Derived] Jenkins AJ, Braffett BH, Basu A, Bebu I, Dagogo-Jack S, Orchard TJ, Wallia A, Lopes-Virella MF, Garvey WT, Lachin JM, Lyons TJ; DCCT/EDIC Research Group. Serum urate and cardiovascular events in the DCCT/EDIC study. Sci Rep. 2021 Jul 9;11(1):14182. doi: 10.1038/s41598-021-90785-4. PMID 34244538
- [Derived] Jacobson AM, Ryan CM, Braffett BH, Gubitosi-Klug RA, Lorenzi GM, Luchsinger JA, Trapani VR, Bebu I, Chaytor N, Hitt SM, Farrell K, Lachin JM; DCCT/EDIC Research Group. Cognitive performance declines in older adults with type 1 diabetes: results from 32 years of follow-up in the DCCT and EDIC Study. Lancet Diabetes Endocrinol. 2021 Jul;9(7):436-445. doi: 10.1016/S2213-8587(21)00086-3. Epub 2021 May 27. PMID 34051936
- [Derived] Gubitosi-Klug R, Gao X, Pop-Busui R, de Boer IH, White N, Aiello LP, Miller R, Palmer J, Tamborlane W, Wallia A, Kosiborod M, Lachin JM, Bebu I; DCCT/EDIC Research Group. Associations of Microvascular Complications With the Risk of Cardiovascular Disease in Type 1 Diabetes. Diabetes Care. 2021 Jul;44(7):1499-1505. doi: 10.2337/dc20-3104. Epub 2021 May 12. PMID 33980605
- [Derived] Bebu I, Keshavarzi S, Gao X, Braffett BH, Canty AJ, Herman WH, Orchard TJ, Dagogo-Jack S, Nathan DM, Lachin JM, Paterson AD; DCCT/EDIC Research Group. Genetic Risk Factors for CVD in Type 1 Diabetes: The DCCT/EDIC Study. Diabetes Care. 2021 Jun;44(6):1309-1316. doi: 10.2337/dc20-2388. Epub 2021 Apr 21. PMID 33883194
- [Derived] Gubitosi-Klug RA, Braffett BH, Hitt S, Arends V, Uschner D, Jones K, Diminick L, Karger AB, Paterson AD, Roshandel D, Marcovina S, Lachin JM, Steffes M, Palmer JP; DCCT/EDIC Research Group. Residual beta cell function in long-term type 1 diabetes associates with reduced incidence of hypoglycemia. J Clin Invest. 2021 Feb 1;131(3):e143011. doi: 10.1172/JCI143011. PMID 33529168
- [Derived] Hainsworth DP, Gao X, Bebu I, Das A, Olmos de Koo L, Barkmeier AJ, Tamborlane W, Lachin JM, Aiello LP; Diabetes Control and Complications Trial and Follow-up Epidemiology of Diabetes Interventions and Complications Research Group. Refractive Error and Retinopathy Outcomes in Type 1 Diabetes: The Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study. Ophthalmology. 2021 Apr;128(4):554-560. doi: 10.1016/j.ophtha.2020.09.014. Epub 2020 Sep 14. PMID 32941962
- [Derived] Bebu I, Braffett BH, Schade D, Sivitz W, Malone JI, Pop-Busui R, Lorenzi GM, Lee P, Trapani VR, Wallia A, Herman WH, Lachin JM; DCCT/EDIC Research Group. An Observational Study of the Equivalence of Age and Duration of Diabetes to Glycemic Control Relative to the Risk of Complications in the Combined Cohorts of the DCCT/EDIC Study. Diabetes Care. 2020 Oct;43(10):2478-2484. doi: 10.2337/dc20-0226. Epub 2020 Aug 11. PMID 32788280
- [Derived] Chen Z, Miao F, Braffett BH, Lachin JM, Zhang L, Wu X, Roshandel D, Carless M, Li XA, Tompkins JD, Kaddis JS, Riggs AD, Paterson AD; DCCT/EDIC Study Group; Natarajan R. DNA methylation mediates development of HbA1c-associated complications in type 1 diabetes. Nat Metab. 2020 Aug;2(8):744-762. doi: 10.1038/s42255-020-0231-8. Epub 2020 Jul 20. PMID 32694834
- [Derived] Braffett BH, Gubitosi-Klug RA, Albers JW, Feldman EL, Martin CL, White NH, Orchard TJ, Lopes-Virella M, Lachin JM, Pop-Busui R; DCCT/EDIC Research Group. Risk Factors for Diabetic Peripheral Neuropathy and Cardiovascular Autonomic Neuropathy in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study. Diabetes. 2020 May;69(5):1000-1010. doi: 10.2337/db19-1046. Epub 2020 Feb 12. PMID 32051148
- [Derived] Bebu I, Schade D, Braffett B, Kosiborod M, Lopes-Virella M, Soliman EZ, Herman WH, Bluemke DA, Wallia A, Orchard T, Lachin JM; DCCT/EDIC Research Group. Risk Factors for First and Subsequent CVD Events in Type 1 Diabetes: The DCCT/EDIC Study. Diabetes Care. 2020 Apr;43(4):867-874. doi: 10.2337/dc19-2292. Epub 2020 Jan 30. PMID 32001614
- [Derived] Braffett BH, Dagogo-Jack S, Bebu I, Sivitz WI, Larkin M, Kolterman O, Lachin JM; DCCT/EDIC Research Group. Response to Comment on Braffett et al. Association of Insulin Dose, Cardiometabolic Risk Factors, and Cardiovascular Disease in Type 1 Diabetes During 30 Years of Follow-up in the DCCT/EDIC Study. Diabetes Care 2019;42:657-664. Diabetes Care. 2019 Aug;42(8):e137. doi: 10.2337/dci19-0026. No abstract available. PMID 31332032
- [Derived] Budoff M, Backlund JC, Bluemke DA, Polak J, Bebu I, Schade D, Strowig S, Raskin P, Lachin JM; DCCT/EDIC Research Group. The Association of Coronary Artery Calcification With Subsequent Incidence of Cardiovascular Disease in Type 1 Diabetes: The DCCT/EDIC Trials. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 2):1341-1349. doi: 10.1016/j.jcmg.2019.01.014. Epub 2019 Mar 13. PMID 30878435
- [Derived] Perkins BA, Bebu I, de Boer IH, Molitch M, Tamborlane W, Lorenzi G, Herman W, White NH, Pop-Busui R, Paterson AD, Orchard T, Cowie C, Lachin JM; Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Research Group. Risk Factors for Kidney Disease in Type 1 Diabetes. Diabetes Care. 2019 May;42(5):883-890. doi: 10.2337/dc18-2062. Epub 2019 Mar 4. PMID 30833370
- [Derived] Hainsworth DP, Bebu I, Aiello LP, Sivitz W, Gubitosi-Klug R, Malone J, White NH, Danis R, Wallia A, Gao X, Barkmeier AJ, Das A, Patel S, Gardner TW, Lachin JM; Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Research Group. Risk Factors for Retinopathy in Type 1 Diabetes: The DCCT/EDIC Study. Diabetes Care. 2019 May;42(5):875-882. doi: 10.2337/dc18-2308. Epub 2019 Mar 4. PMID 30833368
- [Derived] Kim C, Pan Y, Braffett BH, Arends VL, Steffes MW, Wessells H, Sarma AV; DCCT/EDIC Research Group. Anti-Mullerian hormone and its relationships with subclinical cardiovascular disease and renal disease in a longitudinal cohort study of women with type 1 diabetes. Womens Midlife Health. 2017 Aug 18;3:5. doi: 10.1186/s40695-017-0023-9. eCollection 2017. PMID 30766706
- [Derived] Braffett BH, Dagogo-Jack S, Bebu I, Sivitz WI, Larkin M, Kolterman O, Lachin JM; DCCT/EDIC Research Group. Association of Insulin Dose, Cardiometabolic Risk Factors, and Cardiovascular Disease in Type 1 Diabetes During 30 Years of Follow-up in the DCCT/EDIC Study. Diabetes Care. 2019 Apr;42(4):657-664. doi: 10.2337/dc18-1574. Epub 2019 Feb 6. PMID 30728218
- [Derived] Wessells H, Braffett BH, Holt SK, Jacobson AM, Kusek JW, Cowie C, Dunn RL, Sarma AV; DCCT/EDIC Study Group. Burden of Urological Complications in Men and Women With Long-standing Type 1 Diabetes in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Cohort. Diabetes Care. 2018 Oct;41(10):2170-2177. doi: 10.2337/dc18-0255. Epub 2018 Aug 13. PMID 30104298
- [Derived] Herman WH, Braffett BH, Kuo S, Lee JM, Brandle M, Jacobson AM, Prosser LA, Lachin JM. What are the clinical, quality-of-life, and cost consequences of 30 years of excellent vs. poor glycemic control in type 1 diabetes? J Diabetes Complications. 2018 Oct;32(10):911-915. doi: 10.1016/j.jdiacomp.2018.05.007. Epub 2018 Jun 12. PMID 30082172
- [Derived] Herman WH, Braffett BH, Kuo S, Lee JM, Brandle M, Jacobson AM, Prosser LA, Lachin JM. The 30-year cost-effectiveness of alternative strategies to achieve excellent glycemic control in type 1 diabetes: An economic simulation informed by the results of the diabetes control and complications trial/epidemiology of diabetes interventions and complications (DCCT/EDIC). J Diabetes Complications. 2018 Oct;32(10):934-939. doi: 10.1016/j.jdiacomp.2018.06.005. Epub 2018 Jun 12. PMID 30064713
- [Derived] Basu A, Jenkins AJ, Stoner JA, Zhang Y, Klein RL, Lopes-Virella MF, Garvey WT, Schade DS, Wood J, Alaupovic P, Lyons TJ; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Apolipoprotein-defined lipoprotein subclasses, serum apolipoproteins, and carotid intima-media thickness in T1D. J Lipid Res. 2018 May;59(5):872-883. doi: 10.1194/jlr.P080143. Epub 2018 Mar 25. PMID 29576550
- [Derived] de Boer IH, Gao X, Bebu I, Hoofnagle AN, Lachin JM, Paterson A, Perkins BA, Saenger AK, Steffes MW, Zinman B, Molitch ME. Biomarkers of tubulointerstitial damage and function in type 1 diabetes. BMJ Open Diabetes Res Care. 2017 Nov 14;5(1):e000461. doi: 10.1136/bmjdrc-2017-000461. eCollection 2017. PMID 29177052
- [Derived] Purnell JQ, Braffett BH, Zinman B, Gubitosi-Klug RA, Sivitz W, Bantle JP, Ziegler G, Cleary PA, Brunzell JD; DCCT/EDIC Research Group. Impact of Excessive Weight Gain on Cardiovascular Outcomes in Type 1 Diabetes: Results From the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study. Diabetes Care. 2017 Dec;40(12):1756-1762. doi: 10.2337/dc16-2523. PMID 29138273
- [Derived] Bebu I, Braffett BH, Pop-Busui R, Orchard TJ, Nathan DM, Lachin JM; DCCT/EDIC Research Group. The relationship of blood glucose with cardiovascular disease is mediated over time by traditional risk factors in type 1 diabetes: the DCCT/EDIC study. Diabetologia. 2017 Oct;60(10):2084-2091. doi: 10.1007/s00125-017-4374-4. Epub 2017 Jul 16. PMID 28711972
- [Derived] Gubitosi-Klug RA, Braffett BH, White NH, Sherwin RS, Service FJ, Lachin JM, Tamborlane WV; Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Research Group. Risk of Severe Hypoglycemia in Type 1 Diabetes Over 30 Years of Follow-up in the DCCT/EDIC Study. Diabetes Care. 2017 Aug;40(8):1010-1016. doi: 10.2337/dc16-2723. Epub 2017 May 26. PMID 28550194
- [Derived] Lachin JM, Bebu I, Bergenstal RM, Pop-Busui R, Service FJ, Zinman B, Nathan DM; DCCT/EDIC Research Group. Association of Glycemic Variability in Type 1 Diabetes With Progression of Microvascular Outcomes in the Diabetes Control and Complications Trial. Diabetes Care. 2017 Jun;40(6):777-783. doi: 10.2337/dc16-2426. Epub 2017 Apr 12. PMID 28404658
- [Derived] Armstrong AC, Ambale-Venkatesh B, Turkbey E, Donekal S, Chamera E, Backlund JY, Cleary P, Lachin J, Bluemke DA, Lima JA; DCCT/EDIC Research Group. Association of Cardiovascular Risk Factors and Myocardial Fibrosis With Early Cardiac Dysfunction in Type 1 Diabetes: The Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study. Diabetes Care. 2017 Mar;40(3):405-411. doi: 10.2337/dc16-1889. Epub 2016 Dec 16. PMID 27986796
- [Derived] de Boer IH, Gao X, Cleary PA, Bebu I, Lachin JM, Molitch ME, Orchard T, Paterson AD, Perkins BA, Steffes MW, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group. Albuminuria Changes and Cardiovascular and Renal Outcomes in Type 1 Diabetes: The DCCT/EDIC Study. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):1969-1977. doi: 10.2215/CJN.02870316. Epub 2016 Oct 24. PMID 27797889
- [Derived] Writing Group for the DCCT/EDIC Research Group. Coprogression of Cardiovascular Risk Factors in Type 1 Diabetes During 30 Years of Follow-up in the DCCT/EDIC Study. Diabetes Care. 2016 Sep;39(9):1621-30. doi: 10.2337/dc16-0502. Epub 2016 Jul 19. PMID 27436274
- [Derived] Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Study Research Group. Mortality in Type 1 Diabetes in the DCCT/EDIC Versus the General Population. Diabetes Care. 2016 Aug;39(8):1378-83. doi: 10.2337/dc15-2399. Epub 2016 Jul 13. PMID 27411699
- [Derived] Hotaling JM, Sarma AV, Patel DP, Braffett BH, Cleary PA, Feldman E, Herman WH, Martin CL, Jacobson AM, Wessells H, Pop-Busui R; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Cardiovascular Autonomic Neuropathy, Sexual Dysfunction, and Urinary Incontinence in Women With Type 1 Diabetes. Diabetes Care. 2016 Sep;39(9):1587-93. doi: 10.2337/dc16-0059. Epub 2016 Jun 28. PMID 27352953
- [Derived] Roshandel D, Klein R, Klein BE, Wolffenbuttel BH, van der Klauw MM, van Vliet-Ostaptchouk JV, Atzmon G, Ben-Avraham D, Crandall JP, Barzilai N, Bull SB, Canty AJ, Hosseini SM, Hiraki LT, Maynard J, Sell DR, Monnier VM, Cleary PA, Braffett BH; DCCT/EDIC Research Group; Paterson AD. New Locus for Skin Intrinsic Fluorescence in Type 1 Diabetes Also Associated With Blood and Skin Glycated Proteins. Diabetes. 2016 Jul;65(7):2060-71. doi: 10.2337/db15-1484. Epub 2016 Apr 12. PMID 27207532
- [Derived] Lenherr SM, Clemens JQ, Braffett BH, Dunn RL, Cleary PA, Kim C, Herman WH, Hotaling JM, Jacobson AM, Brown JS, Wessells H, Sarma AV; DCCT/EDIC Research Group. Glycaemic control and risk of incident urinary incontinence in women with Type 1 diabetes: results from the Diabetes Control and Complications Trial and Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) study. Diabet Med. 2016 Nov;33(11):1528-1535. doi: 10.1111/dme.13126. Epub 2016 Apr 24. PMID 27028025
- [Derived] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group. Risk Factors for Cardiovascular Disease in Type 1 Diabetes. Diabetes. 2016 May;65(5):1370-9. doi: 10.2337/db15-1517. Epub 2016 Feb 19. PMID 26895792
- [Derived] Sell DR, Sun W, Gao X, Strauch C, Lachin JM, Cleary PA, Genuth S; DCCT/EDIC Research Group; Monnier VM. Skin collagen fluorophore LW-1 versus skin fluorescence as markers for the long-term progression of subclinical macrovascular disease in type 1 diabetes. Cardiovasc Diabetol. 2016 Feb 11;15:30. doi: 10.1186/s12933-016-0343-3. PMID 26864236
- [Derived] Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Study Research Group. Intensive Diabetes Treatment and Cardiovascular Outcomes in Type 1 Diabetes: The DCCT/EDIC Study 30-Year Follow-up. Diabetes Care. 2016 May;39(5):686-93. doi: 10.2337/dc15-1990. Epub 2016 Feb 9. PMID 26861924
- [Derived] Porta M, Toppila I, Sandholm N, Hosseini SM, Forsblom C, Hietala K, Borio L, Harjutsalo V, Klein BE, Klein R, Paterson AD; DCCT/EDIC Research Group; Groop PH; FinnDiane Study Group. Variation in SLC19A3 and Protection From Microvascular Damage in Type 1 Diabetes. Diabetes. 2016 Apr;65(4):1022-30. doi: 10.2337/db15-1247. Epub 2015 Dec 30. PMID 26718501
- [Derived] Kim C, Bebu I, Braffett B, Cleary PA, Arends V, Steffes M, Wessells H, Orchard T, Sarma AV; DCCT/EDIC Research Group. Testosterone and cardiac mass and function in men with type 1 diabetes in the Epidemiology of Diabetes Interventions and Complications Study (EDIC). Clin Endocrinol (Oxf). 2016 May;84(5):693-9. doi: 10.1111/cen.12990. Epub 2016 Jan 25. PMID 26641212
- [Derived] Kim C, Pop-Busui R, Braffett B, Cleary PA, Bebu I, Wessells H, Orchard T, Sarma AV; DCCT/E.D.I.C. Research Group. Testosterone Concentrations and Cardiovascular Autonomic Neuropathy in Men with Type 1 Diabetes in the Epidemiology of Diabetes Interventions and Complications Study (EDIC). J Sex Med. 2015 Nov;12(11):2153-9. doi: 10.1111/jsm.13029. Epub 2015 Nov 12. PMID 26559501
- [Derived] Monnier VM, Sun W, Gao X, Sell DR, Cleary PA, Lachin JM, Genuth S; DCCT/EDIC Research Group. Skin collagen advanced glycation endproducts (AGEs) and the long-term progression of sub-clinical cardiovascular disease in type 1 diabetes. Cardiovasc Diabetol. 2015 Sep 5;14:118. doi: 10.1186/s12933-015-0266-4. PMID 26341632
- [Derived] Eny KM, Orchard TJ, Miller RG, Maynard J, Grant DM, Costacou T, Cleary PA, Braffett BH, Paterson AD; DCCT/EDIC Research Group. Caffeine Consumption Contributes to Skin Intrinsic Fluorescence in Type 1 Diabetes. Diabetes Technol Ther. 2015 Oct;17(10):726-34. doi: 10.1089/dia.2015.0017. Epub 2015 Jul 20. PMID 26192006
- [Derived] Lipska KJ, Montori VM. ACP Journal Club. In type 1 diabetes, intensive insulin therapy for 6.5 y reduced mortality at 27 y compared with usual care. Ann Intern Med. 2015 May 19;162(10):JC12. doi: 10.7326/ACPJC-2015-162-10-012. No abstract available. PMID 25984873
- [Derived] Bharucha AE, Batey-Schaefer B, Cleary PA, Murray JA, Cowie C, Lorenzi G, Driscoll M, Harth J, Larkin M, Christofi M, Bayless M, Wimmergren N, Herman W, Whitehouse F, Jones K, Kruger D, Martin C, Ziegler G, Zinsmeister AR, Nathan DM; Diabetes Control and Complications Trial-Epidemiology of Diabetes Interventions and Complications Research Group. Delayed Gastric Emptying Is Associated With Early and Long-term Hyperglycemia in Type 1 Diabetes Mellitus. Gastroenterology. 2015 Aug;149(2):330-9. doi: 10.1053/j.gastro.2015.05.007. Epub 2015 May 14. PMID 25980755
- [Derived] Pop-Busui R, Hotaling J, Braffett BH, Cleary PA, Dunn RL, Martin CL, Jacobson AM, Wessells H, Sarma AV; DCCT/EDIC Research Group. Cardiovascular autonomic neuropathy, erectile dysfunction and lower urinary tract symptoms in men with type 1 diabetes: findings from the DCCT/EDIC. J Urol. 2015 Jun;193(6):2045-51. doi: 10.1016/j.juro.2014.12.097. Epub 2015 Jan 10. PMID 25584994
- [Derived] Sarma AV, Hotaling J, Dunn RL, Cleary PA, Braffett BH, Kim C, Martin C, Herman W, Gatcomb P, Jacobson AM, Holt SK, Wessells H; DCCT/EDIC Research Group. Poor glycemic control is associated with reduced prostate specific antigen concentrations in men with type 1 diabetes. J Urol. 2015 Mar;193(3):786-93. doi: 10.1016/j.juro.2014.08.115. Epub 2014 Sep 11. PMID 25218922
- [Derived] Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Research Group; Lachin JM, White NH, Hainsworth DP, Sun W, Cleary PA, Nathan DM. Effect of intensive diabetes therapy on the progression of diabetic retinopathy in patients with type 1 diabetes: 18 years of follow-up in the DCCT/EDIC. Diabetes. 2015 Feb;64(2):631-42. doi: 10.2337/db14-0930. Epub 2014 Sep 9. PMID 25204977
- [Derived] DCCT/EDIC research group. Effect of intensive diabetes treatment on albuminuria in type 1 diabetes: long-term follow-up of the Diabetes Control and Complications Trial and Epidemiology of Diabetes Interventions and Complications study. Lancet Diabetes Endocrinol. 2014 Oct;2(10):793-800. doi: 10.1016/S2213-8587(14)70155-X. Epub 2014 Jul 17. PMID 25043685
- [Derived] Eny KM, Lutgers HL, Maynard J, Klein BE, Lee KE, Atzmon G, Monnier VM, van Vliet-Ostaptchouk JV, Graaff R, van der Harst P, Snieder H, van der Klauw MM, Sell DR, Hosseini SM, Cleary PA, Braffett BH, Orchard TJ, Lyons TJ, Howard K, Klein R, Crandall JP, Barzilai N, Milman S, Ben-Avraham D; LifeLines Cohort Study Group; DCCT/EDIC Research Group; Wolffenbuttel BH, Paterson AD. GWAS identifies an NAT2 acetylator status tag single nucleotide polymorphism to be a major locus for skin fluorescence. Diabetologia. 2014 Aug;57(8):1623-34. doi: 10.1007/s00125-014-3286-9. Epub 2014 Jun 17. PMID 24934506
- [Derived] McGee P, Steffes M, Nowicki M, Bayless M, Gubitosi-Klug R, Cleary P, Lachin J, Palmer J; DCCT/EDIC Research Group. Insulin secretion measured by stimulated C-peptide in long-established Type 1 diabetes in the Diabetes Control and Complications Trial (DCCT)/ Epidemiology of Diabetes Interventions and Complications (EDIC) cohort: a pilot study. Diabet Med. 2014 Oct;31(10):1264-8. doi: 10.1111/dme.12504. Epub 2014 Jun 9. PMID 24836354
- [Derived] Larkin ME, Barnie A, Braffett BH, Cleary PA, Diminick L, Harth J, Gatcomb P, Golden E, Lipps J, Lorenzi G, Mahony C, Nathan DM; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Musculoskeletal complications in type 1 diabetes. Diabetes Care. 2014 Jul;37(7):1863-9. doi: 10.2337/dc13-2361. Epub 2014 Apr 10. PMID 24722493
- [Derived] Buschur E, Sarma AV, Pietropaolo M, Dunn RL, Braffett BH, Cleary PA, Cowie C, Larkin ME, Wessells H, Nathan DM, Kim C; DCCT/EDIC Research Group. Self-reported autoimmune disease by sex in the diabetes control and complications trial/epidemiology of diabetes interventions and complications (DCCT/EDIC) study. Diabetes Care. 2014 Feb;37(2):e28-9. doi: 10.2337/dc13-1890. No abstract available. PMID 24459159
- [Derived] de Boer IH, Sun W, Cleary PA, Lachin JM, Molitch ME, Zinman B, Steffes MW; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study Research Group. Longitudinal changes in estimated and measured GFR in type 1 diabetes. J Am Soc Nephrol. 2014 Apr;25(4):810-8. doi: 10.1681/ASN.2013050557. Epub 2013 Dec 5. PMID 24309189
- [Derived] Nathan DM, Bayless M, Cleary P, Genuth S, Gubitosi-Klug R, Lachin JM, Lorenzi G, Zinman B; DCCT/EDIC Research Group. Diabetes control and complications trial/epidemiology of diabetes interventions and complications study at 30 years: advances and contributions. Diabetes. 2013 Dec;62(12):3976-86. doi: 10.2337/db13-1093. No abstract available. PMID 24264395
- [Derived] Kim C, Cleary PA, Cowie CC, Braffett BH, Dunn RL, Larkin ME, Gatcomb PM, Wessells HB, Nathan DM, Sarma AV; DCCT/EDIC Research Group. Effect of glycemic treatment and microvascular complications on menopause in women with type 1 diabetes in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) cohort. Diabetes Care. 2014;37(3):701-8. doi: 10.2337/dc13-1746. Epub 2013 Oct 29. PMID 24170751
- [Derived] Jacobson AM, Braffett BH, Cleary PA, Gubitosi-Klug RA, Larkin ME; DCCT/EDIC Research Group. The long-term effects of type 1 diabetes treatment and complications on health-related quality of life: a 23-year follow-up of the Diabetes Control and Complications/Epidemiology of Diabetes Interventions and Complications cohort. Diabetes Care. 2013 Oct;36(10):3131-8. doi: 10.2337/dc12-2109. Epub 2013 Jul 8. PMID 23835693
- [Derived] Orchard TJ, Lyons TJ, Cleary PA, Braffett BH, Maynard J, Cowie C, Gubitosi-Klug RA, Way J, Anderson K, Barnie A, Villavicencio S; DCCT/EDIC Research Group. The association of skin intrinsic fluorescence with type 1 diabetes complications in the DCCT/EDIC study. Diabetes Care. 2013 Oct;36(10):3146-53. doi: 10.2337/dc12-2661. Epub 2013 Jun 28. PMID 23813757
- [Derived] Orchard TJ, Sun W, Cleary PA, Genuth SM, Lachin JM, McGee P, Paterson AD, Raskin P, Anbinder Y, Levy AP; DCCT/EDIC Research Group. Haptoglobin genotype and the rate of renal function decline in the diabetes control and complications trial/epidemiology of diabetes interventions and complications study. Diabetes. 2013 Sep;62(9):3218-23. doi: 10.2337/db13-0256. Epub 2013 Jun 12. PMID 23761102
- [Derived] Genuth SM, Backlund JY, Bayless M, Bluemke DA, Cleary PA, Crandall J, Lachin JM, Lima JA, Miao C, Turkbey EB; DCCT/EDIC Research Group. Effects of prior intensive versus conventional therapy and history of glycemia on cardiac function in type 1 diabetes in the DCCT/EDIC. Diabetes. 2013 Oct;62(10):3561-9. doi: 10.2337/db12-0546. Epub 2013 Mar 21. PMID 23520132
- [Derived] Turkbey EB, Redheuil A, Backlund JY, Small AC, Cleary PA, Lachin JM, Lima JA, Bluemke DA; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Aortic distensibility in type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2380-7. doi: 10.2337/dc12-0393. Epub 2013 Mar 8. PMID 23474588
- [Derived] Pop-Busui R, Cleary PA, Braffett BH, Martin CL, Herman WH, Low PA, Lima JAC, Bluemke DA; DCCT/EDIC Research Group. Association between cardiovascular autonomic neuropathy and left ventricular dysfunction: DCCT/EDIC study (Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications). J Am Coll Cardiol. 2013 Jan 29;61(4):447-454. doi: 10.1016/j.jacc.2012.10.028. Epub 2012 Dec 19. PMID 23265339
- [Derived] Purnell JQ, Zinman B, Brunzell JD; DCCT/EDIC Research Group. The effect of excess weight gain with intensive diabetes mellitus treatment on cardiovascular disease risk factors and atherosclerosis in type 1 diabetes mellitus: results from the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Study (DCCT/EDIC) study. Circulation. 2013 Jan 15;127(2):180-7. doi: 10.1161/CIRCULATIONAHA.111.077487. Epub 2012 Dec 4. PMID 23212717
- [Derived] Kramer JR, Bayless ML, Lorenzi GM, Ziegler GK, Larkin ME, Lackaye ME, Harth J, Diminick LJ, Anderson KL, Braffett BH, Cleary PA; DCCT/EDIC Study Group. Participant characteristics and study features associated with high retention rates in a longitudinal investigation of type 1 diabetes mellitus. Clin Trials. 2012 Dec;9(6):798-805. doi: 10.1177/1740774512458986. Epub 2012 Oct 1. PMID 23027646
- [Derived] de Boer IH, Sachs MC, Cleary PA, Hoofnagle AN, Lachin JM, Molitch ME, Steffes MW, Sun W, Zinman B, Brunzell JD; Diabetes Control and Complication Trial/Epidemiology of Diabetes Interventions and Complications Study Research Group. Circulating vitamin D metabolites and kidney disease in type 1 diabetes. J Clin Endocrinol Metab. 2012 Dec;97(12):4780-8. doi: 10.1210/jc.2012-2852. Epub 2012 Sep 18. PMID 22990096
- [Derived] Larkin ME, Lorenzi GM, Bayless M, Cleary PA, Barnie A, Golden E, Hitt S, Genuth S. Evolution of the study coordinator role: the 28-year experience in Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC). Clin Trials. 2012 Aug;9(4):418-25. doi: 10.1177/1740774512449532. Epub 2012 Jun 22. PMID 22729476
- [Derived] Turkbey EB, Backlund JY, Genuth S, Jain A, Miao C, Cleary PA, Lachin JM, Nathan DM, van der Geest RJ, Soliman EZ, Liu CY, Lima JA, Bluemke DA; DCCT/EDIC Research Group. Myocardial structure, function, and scar in patients with type 1 diabetes mellitus. Circulation. 2011 Oct 18;124(16):1737-46. doi: 10.1161/CIRCULATIONAHA.111.022327. Epub 2011 Sep 26. PMID 21947298
- [Derived] Gai N, Turkbey EB, Nazarian S, van der Geest RJ, Liu CY, Lima JA, Bluemke DA. T1 mapping of the gadolinium-enhanced myocardium: adjustment for factors affecting interpatient comparison. Magn Reson Med. 2011 May;65(5):1407-15. doi: 10.1002/mrm.22716. Epub 2010 Dec 16. PMID 21500267
- [Derived] Nathan DM, Steffes MW, Sun W, Rynders GP, Lachin JM. Determining stability of stored samples retrospectively: the validation of glycated albumin. Clin Chem. 2011 Feb;57(2):286-90. doi: 10.1373/clinchem.2010.150250. Epub 2010 Oct 28. PMID 21030684
- [Derived] Martin CL, Waberski BH, Pop-Busui R, Cleary PA, Catton S, Albers JW, Feldman EL, Herman WH; DCCT/EDIC Research Group. Vibration perception threshold as a measure of distal symmetrical peripheral neuropathy in type 1 diabetes: results from the DCCT/EDIC study. Diabetes Care. 2010 Dec;33(12):2635-41. doi: 10.2337/dc10-0616. Epub 2010 Sep 10. PMID 20833868
- [Derived] Jacobson AM, Ryan CM, Cleary PA, Waberski BH, Weinger K, Musen G, Dahms W; Diabetes Control and Complications Trial/EDIC Research Group. Biomedical risk factors for decreased cognitive functioning in type 1 diabetes: an 18 year follow-up of the Diabetes Control and Complications Trial (DCCT) cohort. Diabetologia. 2011 Feb;54(2):245-55. doi: 10.1007/s00125-010-1883-9. Epub 2010 Aug 29. PMID 20803190
- [Derived] Larkin ME, Backlund JY, Cleary P, Bayless M, Schaefer B, Canady J, Nathan DM; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group. Disparity in management of diabetes and coronary heart disease risk factors by sex in DCCT/EDIC. Diabet Med. 2010 Apr;27(4):451-8. doi: 10.1111/j.1464-5491.2010.02972.x. PMID 20536518
- [Derived] Younes N, Cleary PA, Steffes MW, de Boer IH, Molitch ME, Rutledge BN, Lachin JM, Dahms W; DCCT/EDIC Research Group. Comparison of urinary albumin-creatinine ratio and albumin excretion rate in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications study. Clin J Am Soc Nephrol. 2010 Jul;5(7):1235-42. doi: 10.2215/CJN.07901109. Epub 2010 May 6. PMID 20448066
- [Derived] Albers JW, Herman WH, Pop-Busui R, Feldman EL, Martin CL, Cleary PA, Waberski BH, Lachin JM; Diabetes Control and Complications Trial /Epidemiology of Diabetes Interventions and Complications Research Group. Effect of prior intensive insulin treatment during the Diabetes Control and Complications Trial (DCCT) on peripheral neuropathy in type 1 diabetes during the Epidemiology of Diabetes Interventions and Complications (EDIC) Study. Diabetes Care. 2010 May;33(5):1090-6. doi: 10.2337/dc09-1941. Epub 2010 Feb 11. PMID 20150297
- [Derived] White NH, Sun W, Cleary PA, Tamborlane WV, Danis RP, Hainsworth DP, Davis MD; DCCT-EDIC Research Group. Effect of prior intensive therapy in type 1 diabetes on 10-year progression of retinopathy in the DCCT/EDIC: comparison of adults and adolescents. Diabetes. 2010 May;59(5):1244-53. doi: 10.2337/db09-1216. Epub 2010 Feb 11. PMID 20150283
- [Derived] Jacobson AM, Paterson AD, Ryan CM, Cleary PA, Waberski BH, Weinger K, Musen G, Dahms W, Bayless M, Silvers N, Harth J, Boright AP; DCCT/EDIC Research Group. The associations of apolipoprotein E and angiotensin-converting enzyme polymorphisms and cognitive function in Type 1 diabetes based on an 18-year follow-up of the DCCT cohort. Diabet Med. 2010 Jan;27(1):15-22. doi: 10.1111/j.1464-5491.2009.02885.x. PMID 20121884
- [Derived] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group; Nathan DM, Zinman B, Cleary PA, Backlund JY, Genuth S, Miller R, Orchard TJ. Modern-day clinical course of type 1 diabetes mellitus after 30 years' duration: the diabetes control and complications trial/epidemiology of diabetes interventions and complications and Pittsburgh epidemiology of diabetes complications experience (1983-2005). Arch Intern Med. 2009 Jul 27;169(14):1307-16. doi: 10.1001/archinternmed.2009.193. PMID 19636033
- [Derived] Musen G, Jacobson AM, Ryan CM, Cleary PA, Waberski BH, Weinger K, Dahms W, Bayless M, Silvers N, Harth J, White N; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Glycemic control and hypoglycemia: is the loser the winner? Response to Perlmuter et al. Diabetes Care. 2009 Apr;32(4):e46; discussion e47. doi: 10.2337/dc08-2264. No abstract available. PMID 19336634
- [Derived] White NH, Sun W, Cleary PA, Danis RP, Davis MD, Hainsworth DP, Hubbard LD, Lachin JM, Nathan DM. Prolonged effect of intensive therapy on the risk of retinopathy complications in patients with type 1 diabetes mellitus: 10 years after the Diabetes Control and Complications Trial. Arch Ophthalmol. 2008 Dec;126(12):1707-15. doi: 10.1001/archopht.126.12.1707. PMID 19064853
- [Derived] Musen G, Jacobson AM, Ryan CM, Cleary PA, Waberski BH, Weinger K, Dahms W, Bayless M, Silvers N, Harth J, White N; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Impact of diabetes and its treatment on cognitive function among adolescents who participated in the Diabetes Control and Complications Trial. Diabetes Care. 2008 Oct;31(10):1933-8. doi: 10.2337/dc08-0607. Epub 2008 Jul 7. PMID 18606979